CLINICAL TRIAL: NCT07170345
Title: Development of a Computer-Aided Diagnosis System for Hepatocellular Carcinoma Microvascular Invasion Based on Preoperative Image Analysis
Brief Title: Computer-Aided Diagnosis for Hepatocellular Carcinoma Microvascular Invasion
Acronym: HCC-MVI-CAD
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Peking Union Medical College Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Beijing YouAn Hospital (Other); Zhujiang Hospital (Other); Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Henan Provincial People's Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Shengjing Hospital (Other); Beijing Tsinghua Changgeng Hospital (Other); Yunnan Cancer Hospital (Other); The First People's Hospital of Yunnan (Other); Guizhou Provincial People's Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); West China Hospital (Other); ZhuHai Hospital (Other); Dazhou Central Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Di Dong, Professor, Chinese Academy of Sciences
Other Study IDs: CASMI008
Record Dates: First submitted 2025-08-28; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma (HCC); Microvascular Invasion (MVI)
Keywords: Hepatocellular Carcinoma; Microvascular Invasion; Computer-Aided Diagnosis System; Artificial Intelligence; Medical Image; Multimodal Model
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We are collecting preoperative multiphase CT images and related clinical information from patients with hepatocellular carcinoma. We plan to include approximately 5,000 retrospective cases and 400 prospective cases. Enrollment will be limited to patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect imaging data, clinical characteristics, and pathological outcomes. No biospecimens will be retained.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (19):
- Peking Union Medical College Hospital: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- First Affiliated Hospital of Kunming Medical University: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- Beijing YouAn Hospital: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- Zhujiang Hospital: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- Meng Chao Hepatobiliary Hospital of Fujian Medical University: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- First Affiliated Hospital of Wenzhou Medical University: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- Fifth Affiliated Hospital, Sun Yat-Sen University: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- Henan Provincial People's Hospital: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- Guangdong Provincial Hospital of Traditional Chinese Medicine: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- Shengjing Hospital: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- Beijing Tsinghua Changgeng Hospital: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- Yunnan Cancer Hospital: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- The First People's Hospital of Yunnan Province: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- Guizhou Provincial People's Hospital: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- First Affiliated Hospital of Guangxi Medical University: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- West China Hospital: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- Zhuhai People's Hospital: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- Dazhou Central Hospital: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC
- Eastern Hepatobiliary Surgery Hospital: patients aged 18 years and older who undergo surgical resection for hepatocellular carcinoma with available pathological evaluation of microvascular invasion. We will collect preoperative multiphase CT images, clinical characteristics, and pathological outcomes.
  Interventions: Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC

INTERVENTIONS:
Diagnostic Test: Computer-Aided Diagnosis System for Preoperative Prediction of MVI in HCC — This intervention is an artificial intelligence-based computer-aided diagnosis (CAD) system developed to predict microvascular invasion (MVI) in patients with hepatocellular carcinoma using preoperative multiphase CT imaging. The system integrates deep learning, radiomics, and expert-defined imaging features to provide risk assessment and visualization of MVI prior to surgery. In this study, the CAD system will be evaluated retrospectively and prospectively in an observational manner only. The results will not influence clinical decision-making or patient management, and all treatments will follow standard of care.

SUMMARY:
Hepatocellular carcinoma (HCC) is a common malignancy in China with a high mortality rate. Its early recurrence and long-term prognosis are closely associated with tumor aggressiveness. Microvascular invasion (MVI), defined as the presence of tumor cells within small branches of the portal or hepatic veins, is a key indicator of malignant biological behavior in HCC. Clinically, MVI is strongly correlated with postoperative early recurrence and serves as an important factor in determining surgical margin extension, adjuvant therapy, and postoperative management strategies.

At present, definitive diagnosis of MVI still relies on postoperative pathological examination, and stable, effective preoperative assessment methods are lacking. Although some studies have attempted to predict MVI using preoperative imaging features, their clinical translation remains limited by poor generalizability, weak interpretability, and insufficient cross-center adaptability.

This study aims to leverage multiphase preoperative CT imaging, artificial intelligence techniques, and clinical prior knowledge to develop a high-performance, generalizable, and interpretable computer-aided diagnostic system for preoperative prediction of HCC-MVI. An observational, prospective evaluation will be conducted to assess system performance and to facilitate the clinical translation of intelligent diagnostic technologies in real-world practice.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a common malignancy in China with a high mortality rate. Early recurrence and long-term prognosis are closely linked to tumor aggressiveness. Microvascular invasion (MVI), defined as the presence of tumor cells within small branches of the portal or hepatic veins, is a critical marker of malignant biological behavior. Clinically, MVI is strongly associated with early postoperative recurrence and serves as an important reference for determining surgical margin extension, adjuvant treatment, and postoperative management strategies. At present, definitive diagnosis of MVI still relies on postoperative pathological examination, and reliable preoperative assessment methods are lacking. Although prior studies have attempted to predict MVI using preoperative imaging, their clinical application remains limited by poor generalizability, weak interpretability, and insufficient cross-center adaptability.

This study aims to develop a high-performance, generalizable, and interpretable computer-aided diagnostic (CAD) system for preoperative prediction of HCC-MVI using multiphase CT imaging, artificial intelligence techniques, and clinical prior knowledge. The system will be evaluated prospectively in an observational, multicenter clinical study to assess its diagnostic value and clinical applicability.

The CAD system integrates three categories of imaging features: (1) high-level representations automatically extracted by deep neural networks; (2) predefined radiomics features such as tumor morphology, texture, and intensity distributions; and (3) structured prior features derived from radiological expertise, including tumor margin blurriness and spatial relationships with adjacent portal veins. Sparse constraints and redundancy suppression mechanisms will be applied to identify stable and efficient MVI-related representations. In addition, the system adopts a spatial domain strategy covering tumor, peritumoral, and distant regions, in order to capture invasion patterns from both local morphology and microenvironmental context, thereby constructing reproducible and clinically interpretable imaging biomarkers.

To overcome the limitations of single-domain models, the system employs a multi-source heterogeneous fusion strategy that integrates morphological-textural features, dynamic enhancement patterns, and spatial graph structures. The model architecture combines convolutional neural networks (CNNs) to capture fine-grained textures, Transformer modules to model long-range dependencies, and graph neural networks (GNNs) to represent tumor-vascular topological relationships. This hybrid approach enables comprehensive understanding of both local details and global structures. Furthermore, the model incorporates uncertainty quantification and attention-like mechanisms to dynamically adjust prediction confidence and generate saliency heatmaps. These outputs are designed to enhance clinicians' interpretability and trust in the system. An interactive visualization interface will also be developed to support risk interpretation and surgical planning.

The study will conduct a prospective observational validation across multiple clinical centers, with unified inclusion/exclusion criteria and standardized data collection protocols. Model predictions will be blindly compared against postoperative pathological results. In addition to conventional metrics (accuracy, sensitivity, specificity, and AUC), the study will observationally evaluate the impact of model-based predictions on preoperative risk stratification and surgical decision-making. By testing the system across diverse patient populations, the study aims to confirm its generalizability, clinical utility, and potential for real-world translation of intelligent diagnostic technologies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Confirmed diagnosis of hepatocellular carcinoma (HCC) according to the Chinese Clinical Practice Guidelines for Primary Liver Cancer.
* Eligible for surgical intervention (hepatic resection or liver transplantation) according to the Chinese Clinical Practice Guidelines for Cancer, including stages Ia, Ib, and IIa.
* Preoperative imaging examination performed within 1 month before surgery.
* Availability of histopathological evaluation with documented microvascular invasion (MVI) status.

Exclusion Criteria:

* History of prior antitumor treatment, including preoperative surgical intervention, transarterial chemoembolization (TACE), radiofrequency ablation (RFA), systemic therapy, or any other preoperative intervention.
* Presence of major vascular invasion, bile duct invasion/thrombosis, extrahepatic metastasis, or lymph node involvement.
* Diffuse hepatocellular carcinoma or tumor rupture with hemorrhage.
* Lack of key data required for primary analysis.
* Poor image quality that prevents reliable qualitative or radiomics analysis.

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of adult patients (≥18 years) with hepatocellular carcinoma who undergo curative-intent surgical treatment, including hepatic resection or liver transplantation, at participating clinical centers. Approximately 5,000 retrospective cases and 400 prospective cases will be included. All participants will have preoperative multiphase CT imaging and postoperative pathological evaluation with documented microvascular invasion (MVI) status.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristic Curve (AUC) | Within 1 month after surgery
  The AUC will be calculated by comparing CAD system predictions with the reference standard of postoperative pathological diagnosis of microvascular invasion in hepatocellular carcinoma.
Accuracy | Within 1 month after surgery
  Accuracy will be defined as the proportion of correctly classified cases (both MVI-positive and MVI-negative) by the CAD system compared with postoperative pathology.

SECONDARY OUTCOMES:
Sensitivity | Within 1 month after surgery
  Sensitivity will be calculated as the proportion of true positive MVI cases correctly identified by the CAD system compared with postoperative pathology.
Specificity | Within 1 month after surgery
  Specificity will be calculated as the proportion of true negative MVI cases correctly identified by the CAD system compared with postoperative pathology.
Calibration | Within 1 month after surgery
  Calibration performance will be assessed using calibration curves, Hosmer-Lemeshow goodness-of-fit tests, and Brier scores, to determine agreement between predicted probabilities and observed MVI outcomes.

OTHER OUTCOMES:
Processing Time | Within 1 month after surgery
  Average computational time required for the CAD system to generate predictions and visualization outputs will be recorded to assess feasibility for integration into clinical workflow.
Physician Confidence Score | Within 1 month after surgery
  Physician Confidence Score will be measured using a questionnaire that asks physicians to rate their confidence in assessing patient risk after reviewing CAD-generated probability scores and saliency maps. Responses will be collected on a 5-point Likert scale (1 = not confident at all, 2 = slightly confident, 3 = moderately confident, 4 = confident, 5 = very confident). The score will be recorded as the numerical Likert scale value selected by each physician.

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Meng Chao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Zhujiang Hospital, Guangzhou, Guangdong
  - Fifth Affiliated Hospital, Sun Yat-Sen University, Zhuhai, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Shengjing Hospital, Shenyang, Liaoning
  - West China Hospital, Chengdu, Sichuan
  - Dazhou Central Hospital, Dazhou, Sichuan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Tsinghua Changgeng Hospital, Beijing
  - Beijing YouAn Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Eastern Hepatobiliary Surgery Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided